CLINICAL TRIAL: NCT00996372
Title: 24-wk Efficacy and Safety of Flibanserin vs Pbo in Naturally Postmenopausal Women in United States
Brief Title: Flibanserin for the Treatment of Hypoactive Sexual Desire Disorder in Postmenopausal Women
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sprout Pharmaceuticals, Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 511.130
Record Dates: First submitted 2009-10-15; First posted 2009-10-16 (Estimated); Results first posted 2014-06-12 (Estimated); Last update posted 2014-06-12 (Estimated); Status verified 2014-05

CONDITIONS: Sexual Dysfunctions, Psychological
MeSH Terms: conditions — Sexual Dysfunctions, Psychological | interventions — flibanserin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- flibanserin 100mg (Experimental): flibanserin 100mg po qd
  Interventions: Drug: flibanserin
- placebo (Placebo Comparator): placebo one tablet po qd
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: flibanserin — patients will be randomized to flibanserin or placebo in a double-blind manner
  Arms: flibanserin 100mg
Drug: placebo — patients will be randomized to flibanserin or placebo in a double-blind manner
  Arms: placebo

SUMMARY:
The objective of this trial is to assess the safety and efficacy of 24-week course of flibanserin for the treatment of Hypoactive Sexual Desire Disorder (HSDD) in naturally postmenopausal women.

ELIGIBILITY:
Inclusion criteria:

* Naturally postmenopausal women of any age with at least one ovary
* Diagnosis of Hypoactive Sexual Desire Disorder, generalized acquired type,of at least six months duration
* Stable, monogamous heterosexual relationship for at least one year
* Willing to discuss sexual issues
* Willing to engage in sexual activity at least once a month
* Normal Pap smear
* Normal mammogram
* Normal uterine lining
* Able to comply with daily use of handheld data entry device

Exclusion criteria:

* Sexual dysfunctions other than HSDD, such as Sexual Aversion Disorder, Substance-induced Sexual Dysfunction, Dyspareunia, Vaginismus, Gender Identity Disorder, Paraphilia and Sexual Dysfunction due to a General Medical Condition
* Partner with inadequately treated organic or psychosexual dysfunction
* Sexual function impaired by psychiatric disorder
* Sexual function impaired by gynecological disorder
* Major Depression
* Suicidal behavior or ideation
* Major life stress that could impair sexual function
* Substance abuse

Min Age: 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 949 (Actual)
Dates: Start 2009-10; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (75):
- United States (75):
  - 511.130.01074 Boehringer Ingelheim Investigational Site, Birmingham, Alabama
  - 511.130.01046 Boehringer Ingelheim Investigational Site, Huntsville, Alabama
  - 511.130.01042 Boehringer Ingelheim Investigational Site, Mobile, Alabama
  - 511.130.01025 Boehringer Ingelheim Investigational Site, Phoenix, Arizona
  - 511.130.01073 Boehringer Ingelheim Investigational Site, Phoenix, Arizona
  - 511.130.01030 Boehringer Ingelheim Investigational Site, Encinitas, California
  - 511.130.01028 Boehringer Ingelheim Investigational Site, Fair Oaks, California
  - 511.130.01037 Boehringer Ingelheim Investigational Site, Irvine, California
  - 511.130.01022 Boehringer Ingelheim Investigational Site, Sacramento, California
  - 511.130.01035 Boehringer Ingelheim Investigational Site, San Diego, California
  - 511.130.01052 Boehringer Ingelheim Investigational Site, San Diego, California
  - 511.130.01016 Boehringer Ingelheim Investigational Site, Torrance, California
  - 511.130.01021 Boehringer Ingelheim Investigational Site, Vista, California
  - 511.130.01051 Boehringer Ingelheim Investigational Site, Westlake Village, California
  - 511.130.01071 Boehringer Ingelheim Investigational Site, Denver, Colorado
  - 511.130.01053 Boehringer Ingelheim Investigational Site, Farmington, Connecticut
  - 511.130.01015 Boehringer Ingelheim Investigational Site, Groton, Connecticut
  - 511.130.01041 Boehringer Ingelheim Investigational Site, New Britain, Connecticut
  - 511.130.01064 Boehringer Ingelheim Investigational Site, Newark, Delaware
  - 511.130.01062 Boehringer Ingelheim Investigational Site, Washington D.C., District of Columbia
  - 511.130.01003 Boehringer Ingelheim Investigational Site, Boynton Beach, Florida
  - 511.130.01056 Boehringer Ingelheim Investigational Site, Clearwater, Florida
  - 511.130.01065 Boehringer Ingelheim Investigational Site, Daytona Beach, Florida
  - 511.130.01020 Boehringer Ingelheim Investigational Site, Miami, Florida
  - 511.130.01024 Boehringer Ingelheim Investigational Site, Miami, Florida
  - 511.130.01070 Boehringer Ingelheim Investigational Site, New Port Richey, Florida
  - 511.130.01043 Boehringer Ingelheim Investigational Site, Orlando, Florida
  - 511.130.01019 Boehringer Ingelheim Investigational Site, St. Petersburg, Florida
  - 511.130.01061 Boehringer Ingelheim Investigational Site, Tampa, Florida
  - 511.130.01066 Boehringer Ingelheim Investigational Site, Tampa, Florida
  - 511.130.01001 Boehringer Ingelheim Investigational Site, West Palm Beach, Florida
  - 511.130.01002 Boehringer Ingelheim Investigational Site, West Palm Beach, Florida
  - 511.130.01009 Boehringer Ingelheim Investigational Site, Atlanta, Georgia
  - 511.130.01023 Boehringer Ingelheim Investigational Site, Atlanta, Georgia
  - 511.130.01008 Boehringer Ingelheim Investigational Site, Sandy Springs, Georgia
  - 511.130.01044 Boehringer Ingelheim Investigational Site, Chicago, Illinois
  - 511.130.01034 Boehringer Ingelheim Investigational Site, Indianapolis, Indiana
  - 511.130.01067 Boehringer Ingelheim Investigational Site, Lafayette, Louisiana
  - 511.130.01013 Boehringer Ingelheim Investigational Site, Baltimore, Maryland
  - 511.130.01031 Boehringer Ingelheim Investigational Site, Bingham Farms, Michigan
  - 511.130.01006 Boehringer Ingelheim Investigational Site, St Louis, Missouri
  - 511.130.01014 Boehringer Ingelheim Investigational Site, Billings, Montana
  - 511.130.01060 Boehringer Ingelheim Investigational Site, Omaha, Nebraska
  - 511.130.01057 Boehringer Ingelheim Investigational Site, Las Vegas, Nevada
  - 511.130.01039 Boehringer Ingelheim Investigational Site, Moorestown, New Jersey
  - 511.130.01017 Boehringer Ingelheim Investigational Site, Endwell, New York
  - 511.130.01047 Boehringer Ingelheim Investigational Site, New Bern, North Carolina
  - 511.130.01027 Boehringer Ingelheim Investigational Site, Winston-Salem, North Carolina
  - 511.130.01033 Boehringer Ingelheim Investigational Site, Cincinnati, Ohio
  - 511.130.01004 Boehringer Ingelheim Investigational Site, Cleveland, Ohio
  - 511.130.01050 Boehringer Ingelheim Investigational Site, Columbus, Ohio
  - 511.130.01059 Boehringer Ingelheim Investigational Site, Columbus, Ohio
  - 511.130.01058 Boehringer Ingelheim Investigational Site, Dayton, Ohio
  - 511.130.01012 Boehringer Ingelheim Investigational Site, Mayfield Heights, Ohio
  - 511.130.01072 Boehringer Ingelheim Investigational Site, Oklahoma City, Oklahoma
  - 511.130.01007 Boehringer Ingelheim Investigational Site, Eugene, Oregon
  - 511.130.01055 Boehringer Ingelheim Investigational Site, Pittsburgh, Pennsylvania
  - 511.130.01048 Boehringer Ingelheim Investigational Site, Columbia, South Carolina
  - 511.130.01068 Boehringer Ingelheim Investigational Site, Mt. Pleasant, South Carolina
  - 511.130.01063 Boehringer Ingelheim Investigational Site, Knoxville, Tennessee
  - 511.130.01010 Boehringer Ingelheim Investigational Site, Nashville, Tennessee
  - 511.130.01036 Boehringer Ingelheim Investigational Site, Nashville, Tennessee
  - 511.130.01018 Boehringer Ingelheim Investigational Site, Corpus Christi, Texas
  - 511.130.01032 Boehringer Ingelheim Investigational Site, Houston, Texas
  - 511.130.01011 Boehringer Ingelheim Investigational Site, Katy, Texas
  - 511.130.01026 Boehringer Ingelheim Investigational Site, San Antonio, Texas
  - 511.130.01005 Boehringer Ingelheim Investigational Site, Salt Lake City, Utah
  - 511.130.01069 Boehringer Ingelheim Investigational Site, Sandy City, Utah
  - 511.130.01040 Boehringer Ingelheim Investigational Site, Norfolk, Virginia
  - 511.130.01049 Boehringer Ingelheim Investigational Site, Norfolk, Virginia
  - 511.130.01029 Boehringer Ingelheim Investigational Site, Richmond, Virginia
  - 511.130.01075 Boehringer Ingelheim Investigational Site, Richmond, Virginia
  - 511.130.01054 Boehringer Ingelheim Investigational Site, Renton, Washington
  - 511.130.01045 Boehringer Ingelheim Investigational Site, Spokane, Washington
  - 511.130.01038 Boehringer Ingelheim Investigational Site, Tacoma, Washington

REFERENCES:
- [Derived] Simon JA, Kingsberg SA, Shumel B, Hanes V, Garcia M Jr, Sand M. Efficacy and safety of flibanserin in postmenopausal women with hypoactive sexual desire disorder: results of the SNOWDROP trial. Menopause. 2014 Jun;21(6):633-40. doi: 10.1097/GME.0000000000000134. PMID 24281236

RESULTS

PARTICIPANT FLOW:
Groups:
- Flibanserin 100mg: flibanserin 100mg po qd
  flibanserin : patients will be randomized to flibanserin or placebo in a double-blind manner
- Placebo: placebo one tablet po qd
  placebo : patients will be randomized to flibanserin or placebo in a double-blind manner
Period: Overall Study
Arm/Group | Flibanserin 100mg | Placebo
Started | 468 | 481
Completed | 365 | 397
Not Completed | 103 | 84

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Flibanserin | Placebo | Total
Number analyzed (Participants) | 468 | 481 | 949
Age, Customized [Number; unit: participants]
  less than 45 years | 8 | 6 | 14
  45-54 years | 192 | 213 | 405
  55-64 | 248 | 237 | 485
  65 years and older | 20 | 25 | 45
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 468 | 481 | 949
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Number; unit: participants]
  White | 398 | 422 | 820
  White Hispanic | 28 | 23 | 51
  Black/African American | 35 | 27 | 62
  Black/African American Hispanic | 0 | 0 | 0
  Asian | 4 | 4 | 8
  Asian Hispanic | 0 | 0 | 0
  American Indian/Alaskan Native | 3 | 4 | 7
  Hawaiian/Pacific Islander | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in the Number of Satisfying Sexual Events
Description: A small handheld electronic device (eDiary) was used by patients to record information about sexual events. Patients were instructed to complete the eDiary every morning. When completing an eDiary entry, patients answered questions regarding their sexual events since their last eDiary entry. If patients missed or were late with their eDiary entry, they could enter information about their sexual events since their most recent entry up to a maximum of seven days in the past.
Time Frame: baseline through 24 weeks
Population: The full analysis set (FAS), consisted of those patients who were randomized to a treatment group, received at least one dose of study medication, had at least one baseline value of either one of the co-primary endpoints or key secondary endpoint, and had data available. The FAS was analyzed for efficacy.
Measure: Mean (Standard Deviation); unit: sexual events
Arm/Group | Flibanserin 100mg | Placebo
Number analyzed (Participants) | 429 | 462
sexual events | 1.0 (2.9) | 0.6 (2.8)

2. Primary Outcome: Change From Baseline in the Score on the Female Sexual Function Index (FSFI) Desire Domain
Description: The FSFI© is a brief, self-administered questionnaire to assess key dimensions of sexual function in women. The scale consists of 19 items that assess sexual function over the past four weeks and yields scores in six domains: desire, arousal, lubrication, orgasm, satisfaction, and pain. The two items in the desire domain are scored from 1 to 5 (with 1 being the lowest report of desire and 5 being the highest). The raw scores of the two items are added together and then multiplied by the domain factor of 0.6. Thus, the score of the desire domain ranges from 1.2 to 6.0 (the higher the score, the higher the reported level of desire).
Time Frame: baseline through 24 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Flibanserin 100mg | Placebo
Number analyzed (Participants) | 432 | 463
units on a scale | 0.7 (0.1) | 0.4 (0.1)

3. Secondary Outcome: Change From Baseline on Question 13 of the Female Sexual Distress Scale Revised (FSDS R)
Description: The FSDS© is a self-administered measure of female personal distress associated with sexual dysfunction. Question 13 inquires about distress specifically related to sexual desire. The range for each question, including Question 13, is 0 (Never) to 4 (Always).
Time Frame: change from baseline to 24 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Flibanserin 100mg | Placebo
Number analyzed (Participants) | 432 | 462
units on a scale | -0.8 (0.1) | -0.6 (0.1)

ADVERSE EVENTS:
Arm/Group | Flibanserin 100mg | Placebo
Serious Adverse Events (participants affected / at risk) | 8/468 | 4/481
Other Adverse Events (participants affected / at risk) | 150/468 | 62/481
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Flibanserin 100mg (N=468) | Placebo (N=481)
diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
ankle fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
wrist fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
dengue fever (Infections and infestations) | 1 (1) | 0 (0)
chronic lymphocytic leukemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
intraventricular hemorrhage (Nervous system disorders) | 1 (1) | 0 (0)
myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0)
pancreatitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
duodenitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
hematemesis (Gastrointestinal disorders) | 1 (1) | 0 (0)
hepatic enzyme increased (Gastrointestinal disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Flibanserin 100mg (N=468) | Placebo (N=481)
dizziness (Nervous system disorders) | 46 (54) | 15 (15)
somnolence (Nervous system disorders) | 41 (44) | 7 (8)
headache (Nervous system disorders) | 28 (29) | 23 (23)
nausea (Gastrointestinal disorders) | 35 (37) | 17 (18)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days